CLINICAL TRIAL: NCT01343849
Title: Blood Test for Breast Cancer Associated Auto Antibodies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eventus Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EventusDx_breast_2011ver2
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; auto antibodies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected Breast cancer subjects

SUMMARY:
Intend of use: A blood test for Cancer Associated Auto Antibodies (CAAA) aimed for better diagnostic management of suspected subjects with breast pathology

Study Description: Blood is collected form patients and serum is tested for the presence of CAAA on experimental test kit.

Objectives: To assess the effectiveness of the CAAA test.

Patient Population: The study population will include any women with suspected breast mass detected by any conventional method, scheduled for biopsy, which will result with a pathological verification of the suspected mass.

Target Population: The target population will be any women with suspected breast mass detected by any conventional method, that today, is scheduled for biopsy.

Structure: Subjects that will be enrolled for the study will be checked for the presence of CAAAb, and the results of the CAAAb test will be compared to the pathology submitted by the physicians in the participating centers.

Sample Size: Total of 1000 samples, of which 620 samples will ensure at least 124 true positive breast cancer subjects verified by biopsy, and 124 true negative breast cancer subjects verified by biopsy. Additional 400 samples will be used for calibrations and training sets.(Multi center study, statistical rationale provided below).

Primary Effectiveness Variables: The effectiveness of the test will be defined by the specificity of the test conditionally that the sensitivity is not lower than a pre-defined level of 95%.

Endpoint: The endpoint of this study is to show that the effectiveness is higher than 50%.

Study Sponsor: Eventus Diagnostics Ltd.

Clinical Monitor: For each site a dedicated CRO will be appointed to monitor the clinical trials. All data will be stored in a protected internet-based database, and any changes of the data will be traced and recorded.

DETAILED DESCRIPTION:
General Information:

Since the mutations of a normal cell that lead to a malignancy, involves changes in the structure and function of the cells, it could be assumed that the immune system has recognized some of these changes as antigenic determinates that should be responded against. For many years, investigators tried to distinguish between cancer patients and healthy population by the difference in specific autoantibodies level. In the healthy population, a baseline of the amount of autoantibodies was determined, and the patient population had to have a statistically significant higher level of autoantibodies. Many examples of this method can be found in the scientific literature [example references - Naora et.al. (2001); mintz et. Al. (2003); Korneeva et. Al (2000)]. The presence of autoantibodies in all population in different levels made it very difficult to find these specifically discriminating antibodies. To date, no specific autoantibody is distinguishing solely between healthy and cancer patients (as opposed to autoimmune diseases, where specific autoantibodies can be found in very high levels in patients only).

Our work assumes that specific Autoantibodies expression level should be altered in cancer, and thus these differences can indicate the presence / absence of cancer.

In this experiment protocol, we are checking for differences in expression levels of specific autoantibodies of suspected breast pathology.

Future CAAA Test Intend of use - Identification of specific breast CAAAs, could provide the clinician with additional immunological and antigenic information regarding the patient's condition or medical status.

Test major steps and components - The CAAA test is comprised of a blood collection and processing step followed by detection of specific auto antibodies with an ELISA based assay and a mathematical processing, with a subsequent classification of the results as "positive" or "negative" for breast cancer.

Study Population:

The study population includes all women that are scheduled for a pathological or cytological confirmation either by any kind of biopsy or cytology, prior to any anti-cancer treatment. The clinical suspicion includes one of the following: positive mammography/US/MRI, and suspected physical check. Final verification ("true positive" or "true negative") will be done in relation to pathology/cytology only.

Subject Selection:

The "true positive" group consists of all sequential patients that satisfy inclusion criteria and have positive biopsy results. The "true negative" group consists of sequential patients that satisfy inclusion criteria and have negative biopsy results.

Written informed consent must be obtained prior to obtaining a blood sample from the patient.

This study will be based on multi-centers participation. The minimum number of sites for the study is 2.

All sites will be within Hospitals either in the surgery department or the relevant specific unit which is responsible for providing care for the BC patients.

The same protocol and the same monitoring routines will be applied to all sites. All CRF data will be submitted electronically through a dedicated and secured internet site, all changes will be tracked. When performing the CAAA tests, the Lab/ Sponsor team will have no information regarding the nature of the sample. This pathological information will be provided for statistical evaluation in parallel to the CAAA test.

STUDY DESIGN:

Overall Description - The current study is a single blind case-control validation study, involving all consecutive breast cancer subjects having positive biopsy results (true positive) and equal number of patients with negative biopsy results (true negative). The purpose of the study is to evaluate the effectiveness of the CAAA test.

The effectiveness of the study is defined as the specificity of the CAAA test for a pre defined sensitivity of 95%.

The study will evaluate the sensitivity of CAAA test to show that it is not below the declared level of 95%.

The study will evaluate the specificity of CAAA test in the new study population.

According to known results of PPV of mammography in various populations we assume that the study population will include about 30% of true positive cancer cases.

As of today, large proportion of the suspected subjects was only diagnosed by final pathology of the biopsy. In this study, the true positive and true negative cases (as verified by biopsy) will be compared to the CAAA test results.

Study Procedures

In the hospital:

First, an identified study subject has to sign an informed consent form, and her Eligibility Form filled ,both should be bar-coded.

Subjects' clinical information acquired from the patient's medical file, including age, medical history and results of tests done leading to the diagnostic evaluation of breast cancer will be recorded on the appropriate, bar-coded, pre-study case report forms. The reports will be electronic via a dedicated and secured internet site, any changes in the database will be recorded and will be traceable. A hard copy of the records will be kept in the department. The study is anonymous and the Department will keep the name of the patient without reveling it to investigators and to the study sponsor.

The doctor/ nurse/ phlebotomist will collect a heparin vacuum tube (about 8ml), label (bar-code) them. The tube with the blood will be packaged in a double sealed container.

The blood will be transported at room temperature (18-25°C), according to the relevant regulations, to the laboratory. Transportation time will be not more than 6 hours.

The blood handling laboratory will collect serum according to the protocol, and the serum will be kept frozen at -80, in properly labeled aliquots. The frozen samples will be sent to the diagnostic laboratory for antibody tests.

In the diagnostic laboratory ELISA based tests for the detection of Auto Antibodies relative expression ratios, will be conducted on each sample according to the lab protocol . The samples will be tested for antibodies levels for the antigens that have been identified on a previous training set. All the data will be permanently recorded directly into a dedicated computer. For each sample all antibody results will be put into the coded patient file. A mathematical algorithm will determine if the sample is positive or negative.

At the Hospital, post biopsy:

2-3 weeks after the biopsy, the CRO will collect from the patient's file the results from the pathology lab and any other relevant information as to the nature of the suspected mass. These results will be recorded on the dedicated and secured internet site and a printed bar-coded CRF will be kept in the Department .

The hospital will preserve slices from the suspected masses (either from biopsy or surgery) for future immuno-histochemical or other studies to be conducted by the sponsor.

The final pathology will be compared with the CAAA test results. The results will be analyzed by a statistician with expertise in cancer population studies.

The patients included in this study are undergoing blood test, and only risks are those involving in blood collection. As treatment is not affected by the results, no risks are subjected to the patients participating in the study.

As the study is being conducted with no link to the individual patient, there is no immediate benefit derived from the additional tests run on the blood sample. Future benefit may be derived from the development of the assay.

The current study is a blind prospective validation study, involving all consecutive suspected breast pathology subjects being scheduled for biopsy during the study duration. The purpose of the study is to assess the sensitivity and specificity of the CAAA test for detection breast cancer in women scheduled for biopsy.

Subjects will be screened for potential participation in the study, according to the inclusion and exclusion criteria.

The data will include parameters of the clinical and pathological state of the subjects and results of CAAA ELISA.

There are two goals of the study.

1. To test that the sensitivity of CAAA is not below the pre-defined level.
2. To evaluate the specificity of CAAA test. Statistical Hypothesis The main condition determining the sample size is to validate that the sensitivity of the test is not lower than the predefined level. The classification rule was established in such a way that the sensitivity in the training set was 100%. We assume that the real sensitivity is not lower that 99%.

Null Hypothesis: The sensitivity of the test is not higher than 95%. Alternative hypothesis: The sensitivity of the test is not less than 99%. Data Management A database management system shall be designed and maintained, including screen preparation, and edit check programming. Pre-entry and post-entry quality control of the clinical data shall be performed at each data entry center. All ELISA test results will be uploaded to the database via an internet based interface, and will be locked against further changes. In order to change ELISA test results, unlocking of the database requires consent from the local CRO, the sponsor and the site physician. Unlocking will be done only by the webmaster, and will be recorder in the tracing system component, and in a hard copy held both by the sponsor and the CRO in the site.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 18 years or over.
* Subjects suspected of breast cancer. The clinical suspicion will include one of the following: positive mammography, ultrasound (US), magnetic resonance imaging (MRI), suspected physical exam. Final analysis will be done in relation to pathology only.
* Subjects scheduled biopsy/surgery

Exclusion Criteria:

* Female Subjects less than 18 years of age
* Previous or concurrent malignancies
* Autoimmune disorders diagnosed subjects
* Hematological malignancies
* Subjects under active chemotherapy treatment or chemotherapy in the past 6 months
* Steroid treatment in the past 3 months
* Subject undergoing immunosuppressive treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes all women that are scheduled for a pathological or cytological confirmation either by any kind of biopsy or cytology, prior to any anti-cancer treatment. The clinical suspicion includes one of the following: positive mammography/US/MRI, and suspected physical check. Final verification ("true positive" or "true negative") will be done in relation to pathology/cytology only.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-09; Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tanir Allweis, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Eventus Diagnostics, Ora, Jerusalem, Israel